CLINICAL TRIAL: NCT07263607
Title: A Multicenter Clinical Study on Taurine Treatment for Multiple Sclerosis
Brief Title: A Multicenter Clinical Trial Evaluating the Efficacy and Safety of Taurine as an Adjunctive Therapy in Multiple Sclerosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Academy of Medical Sciences (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other); Tang-Du Hospital (Other); The First Affiliated Hospital of Hainan Medical College (Unknown); Lanzhou University Second Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Daping Hospital of Army Medical University (Other); Shandong Provincial Hospital (Other Government); Afﬁliated Hospital of North Sichuan Medical College (Other); Beijing Tiantan Hospital (Other); The People's Hospital of Leshan (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-590-1
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis (MS) Relapsing Remitting
Keywords: multiple sclerosis; taurine; multicenter, randomized, open-label clinical trial
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Taurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Taurine + DMTs (Experimental): Experimental group
  Interventions: Drug: DMTs + taurine
- DMTs (Placebo Comparator): control
  Interventions: Drug: DMTs

INTERVENTIONS:
Drug: DMTs + taurine — DMTs + Taurine
  Arms: Taurine + DMTs
Drug: DMTs — DMTs
  Arms: DMTs

SUMMARY:
This multicenter, randomized, open-label clinical trial aims to evaluate the efficacy and safety of taurine as an adjunctive therapy to standard disease-modifying treatments (DMTs) in patients with multiple sclerosis (MS). The study seeks to determine whether oral taurine can reduce the number and volume of new or enlarging MRI lesions, decrease relapse rates, and slow disability progression as measured by the Expanded Disability Status Scale (EDSS). It will also explore the effects of taurine on gut microbiota composition, serum neurodegeneration biomarkers (GFAP and NfL), and cognitive function assessed by MMSE and MoCA. Approximately 80 eligible participants will be enrolled and randomly assigned to either continue standard DMT therapy or receive taurine supplementation in addition to DMTs. The treatment duration will be 24 months, with follow-up visits every 3 months for clinical assessment, blood and stool sample collection, and MRI scans every 6 months. This study aims to provide new clinical evidence supporting taurine as a safe and potentially beneficial adjunctive therapy for multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age and Gender: Male or female participants aged 18 to 65 years.
* 2.Diagnosis: Patients diagnosed with multiple sclerosis (MS) according to the 2017 revised McDonald criteria.
* 3.Treatment Background: Patients receiving stable disease-modifying therapy (DMT) prior to enrollment.
* 4. EDSS score between 1.0 and 5.5 at screening.
* 5. Compliance: Ability and willingness to comply with all study procedures, follow-up visits, and study medication requirements.
* 6.Informed Consent: Participants must provide written informed consent before any study-specific procedures are performed.
* 7 Female participants must be non-pregnant and non-lactating, or, if of childbearing potential, must agree to use effective contraception during the study

Exclusion Criteria:

* 1. Patients with known hypersensitivity to taurine or any of its components
* 2. Women who are pregnant or breastfeeding
* 3. Patients currently participating in other clinical trials
* 4. Patients who refuse to participate in the relevant clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
MRI leision activity | From enrollment to the end of treatment at 2 years
  Change in the number, size, and volume of new or enlarging T2 and Gd-enhancing T1 lesions on brain and spinal MRI scans

SECONDARY OUTCOMES:
EDSS score | From enrollment to the end of treatment at 2 years
  Change in Expanded Disability Status Scale (EDSS) score to assess disability progression or improvement
Annualized Relapse Rate (ARR) | From enrollment to the end of treatment at 2 years
  Number of confirmed clinical relapses per patient-year during the 24-month treatment period
Gut Microbiota Composition | From enrollment to the end of treatment at 2 years
  Alterations in gut microbial diversity and relative abundance of key taxa analyzed by 16S rRNA sequencing of stool samples at baseline, Month 12, and Month 24
Serum Biomarkers (GFAP and NfL) | From enrollment to the end of treatment at 2 years
  Change in serum levels of glial fibrillary acidic protein (GFAP) and neurofilament light chain (NfL) from baseline to Month 24 as indicators of neuroinflammation and axonal injury.

OTHER OUTCOMES:
Safety Outcome Measures | From enrollment to the end of treatment at 2 years
  All adverse events occurring during the study period will be recorded, including their onset time, duration, severity, outcome, and relationship to the study drug (taurine). Serious adverse events will be reported immediately according to GCP requirements.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tian J, Song M, Kaufman DL. Homotaurine limits the spreading of T cell autoreactivity within the CNS and ameliorates disease in a model of multiple sclerosis. Sci Rep. 2021 Mar 8;11(1):5402. doi: 10.1038/s41598-021-84751-3. PMID 33686135